CLINICAL TRIAL: NCT02487706
Title: Removal of Dolutegravir by Hemodialysis in HIV-infected Patients With End-stage Renal Disease
Brief Title: Assessment of Dolutegravir Removed by Hemodialysis in HIV-infected Patients With End-stage Renal Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DTG_HD
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: HIV
Keywords: Hemodialysis; HIV-infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dolutegravir 50mg/day per 5 days (Experimental): Dolutegravir 50mg/day per 5 days
  Interventions: Drug: Dolutegravir

INTERVENTIONS:
Drug: Dolutegravir — Dolutegravir 50mg/day per 5 days

SUMMARY:
Data on the capacity of hemodialysis to remove dolutegravir (DTG) from plasma in patients with end-stage renal disease (ESRD) on hemodialysis (HD) are lacking. If DTG was removed from plasma by HD, it would be possible to have subtherapeutic drug concentrations at the end of HD sessions.

DETAILED DESCRIPTION:
The prevalence of chronic renal disease and end-stage renal disease (ESRD) is increasing in the HIV-positive population. This means that an increasing number of HIV-infected patients will need renal replacement therapy.However, little is known about DTG removal from plasma by HD in patients with ESRD.

Objective: to evaluate the effect of HD on DTG clearance as well as on DTG plasma concentrations at steady state in HIV-infected patients with ESRD undergoing HD.

ELIGIBILITY:
Inclusion Criteria

1. Age 1 years old or older.
2. HIV documented infection (western blot)
3. ESRD undergoing routine hemodialysis
4. Stable antiretroviral treatment (no changes within the prior 2 weeks)
5. Signature of informed consent

Exclusion Criteria:

1. Inadequate adherence to antiretroviral treatment (<90% in the week prior to inclusion).
2. Clinical evidence or suspicion that the patient will not be able to comply with the study protocol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
hemodialysis extraction ratio of dolutegravir | Day 5
hemodialysis clearance of dolutegravir | Day 5

SECONDARY OUTCOMES:
percentage of patients presenting adverse events related to dolutegravir | From Baseline to day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Molto J, Graterol F, Miranda C, Khoo S, Bancu I, Amara A, Bonjoch A, Clotet B. Removal of Dolutegravir by Hemodialysis in HIV-Infected Patients with End-Stage Renal Disease. Antimicrob Agents Chemother. 2016 Mar 25;60(4):2564-6. doi: 10.1128/AAC.03131-15. Print 2016 Apr. PMID 26856824